CLINICAL TRIAL: NCT01480687
Title: Effects of Fish Oil Supplementation on Vascular Structure and Function in Hypertensive Patients With Hypertriglyceridemia
Brief Title: Fish Oil Supplementation and Vascular Function in Hypertensive Patients With Hypertriglyceridemia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitario Pedro Ernesto (Other)
Collaborators: Rio de Janeiro State Research Supporting Foundation (FAPERJ) (Other Government)
Responsible Party: Principal Investigator, Mario Fritsch Neves, MD, PhD, Hospital Universitario Pedro Ernesto
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: FO-1800
Record Dates: First submitted 2011-06-22; First posted 2011-11-29 (Estimated); Last update posted 2011-11-29 (Estimated); Status verified 2011-11

CONDITIONS: Hypertension; Hypertriglyceridemia
Keywords: Hypertension; Endothelial dysfunction; Vascular stiffness
MeSH Terms: conditions — Hypertension; Hypertriglyceridemia | interventions — ciprofibrate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Omega-3 fatty acid (Experimental)
  Interventions: Dietary Supplement: DHA-EPA
- Ciprofibrate (Active Comparator)
  Interventions: Drug: Ciprofibrate

INTERVENTIONS:
Dietary Supplement: DHA-EPA — 1800 mg/day
  Other Names: OMEVITS
  Arms: Omega-3 fatty acid
Drug: Ciprofibrate — 100 mg/day
  Other Names: LIPLESS
  Arms: Ciprofibrate

SUMMARY:
The objective of this study is to compare the effects of ciprofibrate versus omega-3 fatty acid supplementation on the vascular structure and function in hypertensive patients with hypertriglyceridemia.

DETAILED DESCRIPTION:
Hypertensive patients aged 40-65 years, both genders, presenting serum triglycerides levels higher than 150 mg/dl will be randomized into two groups. The first group will be receiving ciprofibrate 100mg/day and the second group will be receiving fish oil 1800mg/day. All patients will be evaluated with brachial flow-mediated dilation and with EndoPAT to assess endothelial function before and after supplementation. SPHYGMOCOR and pulse wave velocity (PWV) measurements will also be obtained.

ELIGIBILITY:
Inclusion Criteria:

* Previous diagnosis of hypertension
* Patients with serum triglycerides levels ≥ 150 mg/dl and <500 mg/dl
* Patients on stable antihypertensive medication for at least 4 weeks
* Patients with food consumption maintained for at least 4 weeks

Exclusion Criteria:

* Smoking
* Secondary hypertension
* Hormone replacement therapy
* Diabetes mellitus
* Chronic kidney disease
* Known coronary artery disease
* Previous stroke
* Dyslipidemia severe, with LDL cholesterol> 160 mg/dL or triglycerides ≥ 500 mg/dl
* Use of statins or beta blockers

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2011-05; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Endothelial function | 3 months
  Endothelial function evaluated by brachial flow-mediated dilation and by peripheral arterial tonometry.

CONTACTS AND LOCATIONS:
Overall Officials: Marcela A Casanova, MSc, Principal Investigator — State University of Rio de Janeiro; Mario F Neves, MD, PhD, Study Chair — State University of Rio de Janeiro; Wille Oigman, MD, PhD, Study Chair — State University of Rio de Janeiro; Fernanda J Medeiros, PhD, Study Chair — Federal University of the State of Rio de Janeiro
Locations (1):
- Hospital Universitario Pedro Ernesto, Rio de Janeiro, RJ, Rio de Janeiro, Brazil